CLINICAL TRIAL: NCT06269419
Title: Observational Cohort Study of Natural Course Progression of Diabetic Retinopathy
Brief Title: Study of Natural Course Progression of Diabetic Retinopathy
Status: Recruiting | Type: Observational
Sponsor: Jie Li (Other)
Responsible Party: Sponsor-Investigator, Jie Li, associate chief physician, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Other Study IDs: 2023-KY295
Record Dates: First submitted 2024-02-06; First posted 2024-02-21 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Biomarkers of Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 diabetes patients with no diabetic retinopathy
- Type 2 diabetes patients with mild to moderate diabetic non-proliferative retinopathy

SUMMARY:
The goal of this observational study is to observe the formation and development of the non-perfusion area of diabetic retinopathy in the posterior area of the retina in type 2 diabetes patients aged 18-75 years old, who can cooperate with all examinations and sign informed consent, clinical myopathy examination and Optos 7 field of vision with mild than severe NPDR, and no other exclusion indicators.The main questions it aims to answer are whether posterior retinal non-perfusion area occurs earlier than peripheral non-perfusion area and whether the rate of non-perfusion area expansion is a risk factor for the progression of diabetic retinopathy.

Participants will have protocol-specific follow-up examinations at 1, 2, 3, 4, and 5 years (± 3 months). Additional visits are made as required by the study and the patient's condition.

The contents of follow-up examinations are:

History of other diseases, medications being used, eye diseases, surgeries, treatments, height, weight, and blood pressure.

Best corrected vision, logarithmic visual acuity chart. Tupai OCTA, 24×20mm range, 6×6mm range scan. Optos fundus imaging, color and no red light images. Fundus fluorescence angiography (only preliminary examination for the first time found mild to moderate NPDR patients, who have been angiographed in the past, only at the 5th year, or as required by the condition).

Glycosylated hemoglobin. Creatinine, urea, glomerular filtration rate. Total cholesterol, triglycerides, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol.

Urinary microalbumin/urinary creatinine ACR. Microvisual field.

ELIGIBILITY:
Inclusion criteria:

* Patients with type 2 diabetes aged 18-75 years
* Can cooperate with the inspection and sign the informed consent
* There are no other eye diseases that cause retinal neovascularization
* There is no known substantial media haze that would hinder fundus image acquisition
* No history of fundus laser treatment or no possibility of laser treatment expected within six months
* No previous history of intravitreal drug injection, and no intravitreal drug injection is expected in the next 6 months
* Macular edema without diabetes (Zeiss OCT women < 290µm, male < 305µm; OCT female in Heidelberg is < 305µm, and for males < 320µm)
* In the field of visual field of clinical mydriasis and Optos photo 7 field of view, DR Lesions were less severe than NPDR
* No history of eye surgery

Exclusion criteria:

* Patients with kidney failure.
* History of systemic anti-VEGF therapy within the last month.
* Follow-up is expected to be difficult or patients from other provinces have traction retinal detachment;
* The patient has a history of allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes patients aged 18-75 years old, who can cooperate with all examinations and sign informed consent, clinical myopathy examination and Optos 7 field of vision with mild than severe NPDR, and no other exclusion indicators.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-25 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Observation and follow-up of biomarkers of diabetic retinopathy | 2024-2029
  The biomarkers of diabetic retinopathy were observed by eye examinations including best corrected visual acuity, logarithmic visual acuity chart, TupaOCTA 24×20mm, 6×6mm scan, Optos fundus color and non-red light images, microvisual field at each follow-up.
Level of Glycosylated hemoglobin | 2024-2029
  tested by venous blood
Creatinine | 2024-2029
  tested by venous blood
Total cholesterol | 2024-2029
  tested by venous blood
Urinary microalbumin | 2024-2029
  tested by urine
Urea | 2024-2029
  tested by venous blood
Glomerular filtration rate | 2024-2029
  tested by venous blood
Triglycerides | 2024-2029
  tested by venous blood
Low-density lipoprotein cholesterol | 2024-2029
  tested by venous blood
High-density lipoprotein cholesterol | 2024-2029
  tested by venous blood
Urinary creatinine ACR | 2024-2029
  tested by urine

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Academy of Medical Science Sichuan Provincial Hosptial, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
2030, via https://pan.baidu.com
Supporting Information: CSR
Time Frame: 2030 and for forever
Access Criteria: https://pan.baidu.com
URL: https://pan.baidu.com